CLINICAL TRIAL: NCT03629509
Title: Implementation of the Begin Exploring Fertility Options, Risks and Expectations (BEFORE) Decision Aid - A Stepped Wedge Cluster Randomized Trial
Brief Title: BEFORE Decision Aid Implementation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Applied Health Research Centre (Other); Canadian Breast Cancer Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Nancy Baxter, Chief of General Surgery, Scientist, Unity Health Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-361
Record Dates: First submitted 2018-08-07; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Decision Support Techniques; Breast Neoplasm Female; Young Adult; Evaluation Studies
Keywords: decision aid; breast cancer; young females; implementation; stepped wedge trial
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Cluster Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-Intervention (Other): The BEFORE decision aid will be available for use on the RUBY communication portals (Twitter, Facebook and study portal)
  Data will be collected 6 weeks before the implementation of the BEFORE decision aid in RUBY sites to establish a baseline
  Interventions: Behavioral: BEFORE decision aid
- BEFORE Decision Aid Intervention (Experimental): Evaluate more intensive strategies to promote use of the BEFORE decision aid through:
  1. We will advertise the availability of the BEFORE decision aid with posters placed in clinic areas at each RUBY site, and will have small handouts available to be distributed in clinic.
  2. We will conduct an educational intervention describing and promoting the use of the BEFORE decision aid and general oncofertility information to nurses and support staff at each RUBY site. This will include an optional 1hr informational webinar, direct outreach and training of nurses/support staff on the use of the tool.
  Interventions: Behavioral: BEFORE decision aid
- Post-Intervention (Other): Data will be collected after the BEFORE decision aid has been implemented in each RUBY site regarding the recommendation of fertility resources, most useful/least useful tool, and use of the BEFORE decision aid.
  Interventions: Behavioral: BEFORE decision aid

INTERVENTIONS:
Behavioral: BEFORE decision aid — Implementation of the BEFORE decision aid in clinical practice
  Arms: BEFORE Decision Aid Intervention
Behavioral: BEFORE decision aid — Implementation of the BEFORE decision aid on RUBY communication portals
  Arms: Pre-Intervention
Behavioral: BEFORE decision aid — Review impact of BEFORE decision aid implementation in clinical practice
  Arms: Post-Intervention

SUMMARY:
Fertility is of great importance to young women with cancer. Concerns about the ability to become pregnant after cancer treatment may influence treatment decisions and fertility decision-making is challenging. Despite these challenges, there is a lack of fertility decision support tools. Our team developed the Begin Exploring Fertility Options, Risks and Expectations (BEFORE) decision aid for young breast cancer patients in Canada. This study aims to evaluate the implementation of the BEFORE decision aid in hospital settings through a stepped wedge cluster randomized trial.

DETAILED DESCRIPTION:
The investigators will conduct a stepped wedge cluster randomized trial to sequentially implement the BEFORE decision aid in clinical settings that are currently recruiting young breast cancer patients for the Reducing the bUrden of Breast cancer in Young women (RUBY) Study (www.womensresearch.ca/ruby-study/).

For this trial 24 participating RUBY sites were grouped into 14 clusters (1 to 3 sites per cluster). The decision aid intervention will be sequentially rolled out over the course of 48 weeks to all clusters. None of the clusters will be switched from control to intervention during the first 6 weeks of the study to establish a baseline. Then two clusters will move from the control to the intervention every 6 weeks (called a 'step'). There will be 7 steps total during the study period. At the end of the 7th step all clusters (i.e., participating RUBY sites) will have received the decision aid intervention. The time-point of when the clusters will be switched from control to intervention will be randomized.

The data collection includes obtaining secondary data collected as part of the RUBY study from all patient participants who were enrolled in RUBY during the study period. The primary outcome is the number of patients reporting that fertility tools were recommended to them, based on RUBY participant responses to a 3-month fertility questionnaire. The investigators hypothesizes that following the implementation of the decision aid intervention a 20% difference will be observed, from 10% in the control to 30% in the intervention, in the number of patients who report that someone in their care team recommended a fertility tool.

ELIGIBILITY:
Inclusion Criteria:

* Young females diagnosed with histologically-confirmed breast cancer will be eligible to participate if they:

  1. are age =18 years and prior to their 41st birthday;
  2. are able to provide verbal informed consent and complete the interviews in English or French;
  3. completed the 3-month fertility questionnaire as part of the RUBY Study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 224 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-reported outcome questionnaire - Fertility Preservation Questionnaire | 3 months from date of randomization
  Number of patients reporting that fertility tools were recommended to them following their breast cancer diagnosis

SECONDARY OUTCOMES:
BEFORE decision aid online survey - Provider Recommendation of Decision Aid | From date of randomization until the end of the study at 48 weeks
  Specific provider who recommended the BEFORE decision aid to the patient
BEFORE decision aid online survey - Patient Learning About Decision Aid | From date of randomization until the end of the study at 48 weeks
  How the patient first learned about the aid (e.g, by the poster or their care provider)
BEFORE decision aid online survey - Patient Satisfaction | From date of randomization until the end of the study at 48 weeks
  Patient satisfaction with the way they found out about the BEFORE decision aid

OTHER OUTCOMES:
Google Analytics - Number of Visits | From date of randomization until the end of the study at 48 weeks
  Number of visits to the BEFORE decision aid
Google Analytics - Length of Visits | From date of randomization until the end of the study at 48 weeks
  Length of visits to the BEFORE decision aid
Google Analytics - Most Visited Page | From date of randomization until the end of the study at 48 weeks
  Most visited page on the BEFORE decision aid
Google Analytics - Least Visited Page | From date of randomization until the end of the study at 48 weeks
  Least visited page on the BEFORE decision aid
Google Analytics - Decision Aid Download | From date of randomization until the end of the study at 48 weeks
  Number of people who downloaded the paper BEFORE decision aid
Google Analytics - User Location | From date of randomization until the end of the study at 48 weeks
  BEFORE decision aid user location by province in Canada

CONTACTS AND LOCATIONS:
Overall Officials: Nancy N Baxter, MD, FRCSC, FACS, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: BEFORE decision aid — https://fertilityaid.rethinkbreastcancer.com